CLINICAL TRIAL: NCT04485351
Title: Assessing the Impact of the COVID-19 Lockdown on Metabolic Control and Access to Health Care in Patients With Diabetes: a Monocentric Cross-sectional Study
Brief Title: Assessing the Impact of the COVID-19 Lockdown on Metabolic Control and Access to Health Care in Patients With Diabetes
Acronym: CONFI-DIAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI137
Record Dates: First submitted 2020-07-02; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus; Coronavirus Infection; Metabolic Disease; Glucose Metabolism Disorders
Keywords: diabetes mellitus; lockdown; covid-19
MeSH Terms: conditions — Diabetes Mellitus; Coronavirus Infections; Metabolic Diseases; Glucose Metabolism Disorders; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients from the University Hospital of Nancy
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The outbreak of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and the COVID-19 (Coronavirus Disease-2019) in December 2019 has led to an unprecedented international health situation. Exceptional measures have been taken by public authorities worldwide in order to slow the spread of the virus and prevent healthcare systems from becoming overloaded. In France, a national lockdown has been established during approximately 2 months to increase social distancing and restrict population movements. Hospital routine care appointments have been cancelled, in order to reallocate medical resources towards COVID-19 units and limit contacts between patients within hospitals or waiting rooms. While the virus itself, the disease and potential treatments are currently extensively studied, little data are available on the effect of these public health decisions on the management of a chronic condition such as diabetes.

The French regional CONFI-DIAB study aims at assessing the collateral impact of routine care cancellation during the national lockdown due to COVID-19 in patients with a chronic condition such as diabetes. Special attention will be given to metabolic control and access to health care.

This cross-sectional study should provide information on the consequences of a global lockdown and the associated routine care cancellation on the management of diabetes, and inform future decision making in the event of a new pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patient with diabetes known for at least 6 months before inclusion
* Patient followed by a specialist physician from the University Hospital of Nancy for routine care within the 6 months prior to the lockdown.
* Patient who was assessed for prioritization of care following the end of the lockdown by the department of endocrinology, diabetology and nutrition

Exclusion Criteria:

* Subjects opposed to the use of their data
* Minors, adults under guardianship, protected persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients routinely followed by a specialist physician from the University Hospital of Nancy for diabetes
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Compare glycated hemoglobin levels of patients with diabetes from the University Hospital of Nancy between the period preceding and following the lockdown related to the COVID-19 pandemic. | 6 months period prior to lockdown - 6 weeks period following the end of the lockdown
  HbA1c levels before and after the lockdown period. A 3 months period is required between the 2 values.

SECONDARY OUTCOMES:
Describe the clinical and biological characteristics of patients with diabetes followed in routine care at the University Hospital of Nancy | 6 weeks period following the end of the lockdown
  Use type of diabetes, BMI, lipid profile, micro- and macro-comorbidities and usual therapies from medical records
Describe the change from baseline of biological and clinical parameters of patients with diabetes followed in routine care at the University Hospital of Nancy between the period preceding and following the lockdown. | 6 months period prior to lockdown - 6 weeks period following the end of the lockdown
  Use BMI, lipid profile, renal and hepatic function from medical records
Describe the proportion of patients who presented with one or more significant clinical event during the lockdown. | 6 weeks period following the end of the lockdown
  Ketosis, Ketoacidosis, severe hypoglycemia, COVID-19 infection, hospitalization
Describe the proportion of patients who forgot and/or discontinued one or several medication(s) during the lockdown. | 6 weeks period following the end of the lockdown
  Proportion of patients who forgot and/or discontinued one or several medication(s), medication involved, duration and frequency of omission/discontinuation
Describe the proportion of patients who changed their lifestyle's habits during the lockdown. | 6 weeks period following the end of the lockdown
  Porportion of patients who modified their usual level of physical activity and/or their consumption of alcohol and/or tobacco
Describe healthcare consumption of patients with diabetes during the lockdown. | 6 weeks period following the end of the lockdown
  Proportion of patients who consulted their GP, a specialist physician, pharmacist, biologist, nurse, paramedic, other healthcare professional; type of visit (regular face to face, telemedecine); method for prescription renewal; reason for delay in care; hospitalization (excluding for COVID-19)
Describe the proportion of patients who (1) was tested for SARS-CoV-2 by PCR, (2) developped COVID-19 confirmed by PCR and (3) was hospitalized due to the severity of COVID-19. | 6 weeks period following the end of the lockdown
  Proportion of patients who (1) was tested for SARS-CoV-2 by PCR, (2) developped COVID-19 confirmed by PCR and (3) was hospitalized due to the severity of COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Ludwig, Dr, Principal Investigator — PA
Locations (1):
- University Regional Hospital of Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ludwig L, Scheyer N, Remen T, Guerci B. The Impact of COVID-19 Lockdown on Metabolic Control and Access to Healthcare in People with Diabetes: the CONFI-DIAB Cross-Sectional Study. Diabetes Ther. 2021 Aug;12(8):2207-2221. doi: 10.1007/s13300-021-01105-y. Epub 2021 Jul 9. PMID 34241812